CLINICAL TRIAL: NCT00033371
Title: A Two-Arm Phase II Chemoprevention Trial in Adenomatous Polyposis Coli Patients
Brief Title: Celecoxib With or Without Eflornithine in Preventing Colorectal Cancer in Patients With Familial Adenomatous Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00844; NCI-2013-00844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN95040; CDR0000069278; NCI-P02-0219; ID00-109 (Other: MD Anderson Cancer Center); P30CA016672 (NIH); MDA-ID-00109 (Other: MD Anderson Cancer Network); N01-CN-95040 (Other: DCP); N01CN95040 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer; Familial Adenomatous Polyposis
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyposis Coli | interventions — Celecoxib; Eflornithine; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Celecoxib and Placebo (Active Comparator): Celecoxib 400 mg orally twice daily (PO BID) and Placebo once a day. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Celecoxib; Other: Placebo; Other: Laboratory biomarker analysis; Other: Questionnaire administration
- Arm II: Celecoxib and Eflornithine (Experimental): Celecoxib 400 mg PO BID and Eflornithine PO daily 0.5 g/m^2/day rounded down to the nearest 250 mg dose. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Celecoxib; Drug: eflornithine; Other: Laboratory biomarker analysis; Other: Questionnaire administration

INTERVENTIONS:
Drug: Celecoxib — Given 400 mg PO twice a day
  Other Names: Celebrex; SC-58635
Other: Placebo — Given PO to match DFMO
  Other Names: PLCB
  Arms: Arm I: Celecoxib and Placebo
Drug: eflornithine — Given PO at 0.5 gm/m^2/day rounded down to the nearest 250 mg dose (BSA of < 1.4 = 500 mg/day; BSA of 1.5 - 2.0 = 750 mg/day; BSA of 2.1 - 2.5 = 1000 mg/day; BSA of > 2.6 = 1,250 mg/day).
  Other Names: 2-difluoromethylornithine; DFMO; difluromethylornithine
  Arms: Arm II: Celecoxib and Eflornithine
Other: Laboratory biomarker analysis — Correlative studies
Other: Questionnaire administration — Ancillary studies
  Other Names: Survey

SUMMARY:
This randomized phase II trial studies how well giving celecoxib with or without eflornithine works in preventing colorectal cancer in patients with familial adenomatous polyposis. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of celecoxib and eflornithine may keep cancer from forming in patients with familial adenomatous polyposis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relative efficacy of celecoxib plus eflornithine (DFMO) versus celecoxib plus DFMO placebo in participants with familial adenomatous polyposis (FAP), as evidenced by the percent change from baseline in the number of polyps in focal area(s) of the colorectum in participants having 5 or more >= 2mm colorectal polyps with or without duodenal polyps at baseline.

II. To determine the relative tolerability and safety of celecoxib + DFMO in FAP study participants.

SECONDARY OBJECTIVES:

I. To determine the percent change in polyp size in focal area(s) of the colorectum II. To determine the change in global colorectal polyp burden III. To determine the percent change in the area of plaque-like duodenal polyps in participants presenting with duodenal disease at baseline.

IV. To analyze the effects of these agents on the following panel of mucosal biomarkers: antigen identified by monoclonal antibody Ki-67 (Ki-67), mitotic index (number and spatial distribution of mitoses), phosphorylated histone H3, cyclin-dependent kinase inhibitor 1A (p21/WAF1/Cip1), apoptosis (Terminal deoxynucleotidyl transferase dUTP nick end labeling [TUNEL]), apoptotic index, BCL2-associated X protein (Bax), B-cell CLL/lymphoma 2 (Bcl-2) and measurement of drug effects in colonic polyp and normal tissue cyclooxygenase (cyclooxygenase-1 [COX-1], cyclooxygenase-2 [COX-2]) protein levels, prostaglandin E2 (PGE2), ornithine decarboxylase and polyamines.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive celecoxib orally (PO) twice daily (BID) and placebo PO daily.

ARM II: Patients receive celecoxib PO BID and eflornithine PO daily.

In both arms, treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of just treatment, patients are followed up at 1-2 months.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION INCLUSION CRITERIA:
* Diagnosis of FAP based on any of the following will be acceptable:

  * > 100 polyps or
  * > 10 polyps and age < 40 years, or > 25 polyps and age > 40 years and characteristic family history (autosomal dominant pattern) including:

    * > 100 polyps in a first degree family member or
    * > 25 polyps in two relatives in two generations, including a first degree family member or
    * Genetic diagnosis in a relative or
  * Genetic diagnosis by in vitro synthesized protein (IVSP) or similar assay
* Willingness to abstain from use of nonsteroidal anti-inflammatory drugs (NSAIDs), including aspirin, for the duration of the study; a cardio-protective dose of aspirin (>= 80 mg) may be permitted but must be reviewed/approved by principal investigator (PI)
* If participant is female and of child bearing potential, she agrees to participate in this study by providing written informed consent, has been using adequate contraception (e.g. abstinence, condom, intrauterine device [IUD], birth control pill, diaphragm and spermicide gel combination) since her last menses and will use adequate contraception during the study, is not lactating, and agrees to undergo a serum pregnancy test at baseline, month 3 and month 6; sexually active males must agree to use an accepted and effective method of contraception
* Colon polyp status: the participant has an endoscopically assessable colonic and/or rectal segment
* Participant has no clinically significant hearing loss that is defined by the patient reporting that their hearing loss affects their everyday life and/or wears a hearing aide
* Participants whose air conduction pure tone audiogram reveals a deficit that differs from the age specific norm by less than 30 dB when averaged across two contiguous test frequencies in either ear are eligible, as long as no self-reported hearing deficit or tinnitus is present
* Willingness and ability to sign informed consent
* RANDOMIZATION INCLUSION CRITERIA:
* The individual has assessable colonic polyps remaining in the colon or rectum post baseline colonoscopy or flexible sigmoidoscopy
* Potential participants must have the following colonic or rectal polyp burden at the conclusion of the baseline endoscopy:

  * Rectum:

    * Five or more polyps >= 2 mm diameter
  * Colon:

    * Five or more polyps >= 2 mm diameter including:

      * Three quantifiable polyps > 3 mm diameter, or two quantifiable polyps > 5 mm diameter
      * In the colon, quantifiable polyps are defined as being within a composite "cloverleaf" photograph that includes a tattoo, the appendix, or the ileocecal valve

Exclusion Criteria:

* REGISTRATION EXCLUSION CRITERIA:
* Anticipated colectomy within eight months of randomization
* History of hypersensitivity to COX-2 inhibitors, sulfonamides, NSAIDs or salicylates
* Chronic use of NSAIDs, including aspirin or Celebrex, at any dose during the six months prior to study entry will require a three-month washout period prior to eligibility beginning with the time of the patient's last dose; participants must voluntarily agree to be off all NSAIDs for three months prior to study enrollment; a cardio-protective dose of aspirin (>= 80 mg) may be permitted but must be reviewed/approved by PI
* The use of fluconazole, lithium or chronic use of adrenocorticosteroids
* History in the past year of discrete gastric or duodenal ulcer of size > 5 mm, except that those with a history of Helicobacter pylori related peptic ulcer disease will become eligible for study upon successfully completing antibiotic treatment of Helicobacter pylori
* History of invasive carcinoma in the past five years other than resected Duke's A/B1 colon cancer or resected non-melanomatous skin cancer
* Partial or complete colectomy within 12 months prior to enrollment
* Inability to return for follow-up tests
* Significant medical or psychiatric problems, (including significant renal, hepatic or hematologic dysfunction) which would make the individual a poor protocol candidate
* Use of any investigational agent within the last 3 months, or at the discretion of the medical monitor
* History of pelvic radiation
* RANDOMIZATION EXCLUSION CRITERIA:
* Anticipated colectomy within eight months of randomization; the results of the initial endoscopies, including pathology reports and blood tests will be reviewed by the study endoscopist and surgeon prior to initiation of drug treatment to determine if the patient can remain on study
* Discrete gastric or duodenal ulcer of size > 5 mm; patients with Helicobacter pylori related peptic ulcers of > 5 mm at the time of the baseline endoscopy will become eligible upon endoscopically documented successful treatment of Helicobacter pylori and of the ulcer(s).
* Hemoglobin (Hgb) < 10.0 gm/dl
* Platelet count < 100,000/ml
* White blood cell (WBC) with differential < 3,000/ml
* Serum glutamate pyruvate transaminase (SGPT) > 1.5 x upper limit of normal, serum glutamic oxaloacetic transaminase (SGOT) > 1.5 upper limit of normal
* Alkaline phosphatase > 1.5 x upper limit of normal
* Bilirubin > 2 x upper limit of normal
* Creatinine > 1.5 x upper limit of normal
* Has had a positive serum pregnancy test within 14 days prior to baseline randomization
* Known or prior coagulopathy
* Elevated C-reactive protein (CRP) (> 3.0 mg/L)
* History of cardiovascular diseases or risk factors that might include one of the following: myocardial infarction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery
* Uncontrolled hypertension (> 135/> 85 mm Hg on three repeated measurements during the 6 weeks prior to enrollment on the study); this pertains to subjects with known diagnosis of hypertension; such subjects will have been invited to participate in the trial following successful treatment of their known hypertension; subjects with diagnosis of hypertension established at study entry will be considered cases of potential "white coat" hypertension; such subjects will be otherwise evaluated for protocol and randomized if they agree to be monitored for blood pressure (BP); if BP remains persistently elevated, subjects will be allowed to remain on-study for three months while undergoing antihypertensive therapy and monitoring; if, at the end of 3 months, subjects cannot demonstrate successful BP control as measured and documented locally, dosing will be suspended; such subjects will nevertheless be urged to complete 6-month off study evaluation, for intention to treat analysis
* Family history of premature coronary disease (i.e. onset < 55 years of age)
* Uncontrolled diabetes; subjects with preexisting diagnosis of diabetes will be eligible to participate in the trial if able to document acceptable management by their treating physician; subjects with diagnosis of diabetes established at study entry will be considered cases of new onset disease; such subjects will be otherwise evaluated for protocol and randomized if they agree to blood sugar monitoring; if glucose remains persistently elevated, subjects will be allowed to remain on-study for three months while undergoing therapy and monitoring; of, at the end of 3 months, subjects cannot demonstrate successful glucose control as measured and documented locally, dosing will be suspended; such subjects will nevertheless be urged to complete 6-month off study evaluation, for intention to treat analysis
* Uncontrolled hypercholesteremia (low-density lipoprotein cholesterol [LDL-C] > 130); hypercholesteremia needs to be controlled following the updated National Cholesterol Education Program Adult Treatment Panel III Guidelines for at least 3 months prior to enrollment on the study; hypercholesteremia treatment should continue during the entire period of Celecoxib treatment on the protocol; this pertains to subjects with known diagnosis of hypercholesterolemia; such subjects will have been invited to participate in the trial following successful treatment of their elevated cholesterol; subjects with diagnosis of hypercholesterolemia established at study entry will be considered cases of new onset disease; such subjects will be otherwise evaluated for protocol and randomized if they agree to cholesterol treatment and monitoring; subjects will be allowed to remain on-study for three months while undergoing therapy and monitoring; if, at the end of 3 months, subjects cannot demonstrate successful cholesterol control as measured and documented locally, dosing will be suspended; such subjects will nevertheless be urged to complete 6-month off study evaluation, for intention to treat analysis
* Metabolic syndrome diagnosis; the diagnosis of metabolic syndrome is made when three or more of these risk factors are present:

  * Waist circumference: Men > 102 cm (> 40 in.); women > 88 cm (> 35 in.)
  * Triglycerides > 150 mg/dl ( > 1.69 mmol/L)
  * High-density lipoprotein cholesterol (HDL-C): Men < 40 mg/dl (< 1.03 mmol/L), women < 50 mg/dl (< 1.29 mmol/L)
  * Blood pressure > 130/85 mm Hg
  * Fasting glucose > 110 mg/dl (> 6.1 mmol/L)
* History of deep venous thrombosis, pulmonary embolism, systemic lupus erythematous, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, Factor V Leiden deficiencies or high homocysteine levels
* Any indications for acetylsalicylic acid (ASA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2001-12-13 (Actual); Primary Completion 2009-02-24 (Actual); Study Completion 2009-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lynch, Principal Investigator — MD Anderson Cancer Network
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lynch PM, Burke CA, Phillips R, Morris JS, Slack R, Wang X, Liu J, Patterson S, Sinicrope FA, Rodriguez-Bigas MA, Half E, Bulow S, Latchford A, Clark S, Ross WA, Malone B, Hasson H, Richmond E, Hawk E. An international randomised trial of celecoxib versus celecoxib plus difluoromethylornithine in patients with familial adenomatous polyposis. Gut. 2016 Feb;65(2):286-95. doi: 10.1136/gutjnl-2014-307235. Epub 2015 Mar 19. PMID 25792707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 13, 2001 to October 21, 2008. All recruitment done in medical clinics, with the trial conducted at the University of Texas MD Anderson Cancer, the Cleveland Clinic in Cleveland and St. Mark's Hospital in Harrow, UK.
Pre-assignment Details: Of the 205 participants with familial adenomatous polyposis (FAP) recruited, 112 were randomized. The study was closed due to slow recruitment with enrollment target almost met.
Groups:
- Arm I: Celecoxib and Placebo: Celecoxib 400 mg orally twice daily (PO BID) and Placebo once a day. Treatment continues for 6 months (up to 200 days).
- Arm II: Celecoxib and Eflornithine: Celecoxib 400 mg PO BID and Eflornithine PO daily 0.5 g/m^2/day rounded down to the nearest 250 mg dose (body surface area (BSA) of < 1.4 = 500 mg/day; BSA of 1.5 - 2.0 = 750 mg/day; BSA of 2.1 - 2.5 = 1000 mg/day; BSA of > 2.6 = 1,250 mg/day). Treatment continues for 6 months (up to 200 days).
Period: Overall Study
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Started | 55 | 57
Completed | 49 | 47
Not Completed | 6 | 10
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: According to the protocol, a patient needed to receive at least 80% of intended overall dose AND at least 80% dose during the final 60 days of the study to qualify as evaluable. One participant was randomized to Arm II but withdrew prior to receiving any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Median (Full Range); unit: years] | 38 [18 to 63] | 38 [19 to 59] | 38 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 46 | 50 | 96
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 53 | 53 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 42 | 43 | 85
  United Kingdom | 13 | 14 | 27
Basis of FAP Diagnosis [Number; unit: participants] — Eligible participants aged 18-65 years required to have clinical diagnosis of FAP based on personal history of one of following a)>100 adenomas; b)>10 adenomas before age 40 years; c)>25 adenomas and, if age>40 years, a characteristic family history (autosomal dominant pattern) including >100 polyps in first degree family member, >25 polyps in 2 relatives in two generations, genetic diagnosis in a relative, or d) genetic diagnosis by sequencing/similar assay. Participants required to have an evaluable colon and/or rectal segment, and 5 or more colorectal polyps' ≥2mm at baseline examination.
  participants
    >100 Polyps | 21 | 23 | 44
    >10 Polyps and age <40 | 28 | 23 | 51
    >25 Polyps and age >40 | 6 | 11 | 17
Colon versus Rectum [Number; unit: participants] — Number of participants with intact colon (Colon); or those with rectum only (Rectum Only).
  participants
    Colon | 19 | 27 | 46
    Rectum Only | 36 | 30 | 66
Number of Landmark Polyps at Baseline Screen [Number; unit: participants]
  0-1 | 3 | 5 | 8
  2-4 | 7 | 12 | 19
  5-9 | 19 | 21 | 40
  10 or more | 22 | 19 | 41
  No Baseline Screen | 4 | 0 | 4
Number of Landmark Polyps at least 2 mm at Baseline Screen [Number; unit: participants]
  0-1 | 13 | 20 | 33
  2-4 | 12 | 23 | 35
  5-9 | 22 | 8 | 30
  10 or more | 4 | 6 | 10
  No Baseline Screen | 4 | 0 | 4
Number Landmark Polyps at least 2 mm at Baseline Screen for Evaluable polyps, Evaluable Participants [Number; unit: participants]
  0-1 | 9 | 13 | 22
  2-4 | 11 | 13 | 24
  5-9 | 13 | 5 | 18
  10 or more | 0 | 4 | 4
  No Baseline Screen | 4 | 0 | 4
  Not Evaulable Participant | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Number of Polyps Greater Than or Equal to 2mm in Diameter in Focal Area(s) of the Colorectum
Description: Differences between average treatment effects of two study arms tested using two-sided type I error rate of 5% in two-sample t-test. If model assumptions not met by data or transformations of data, appropriate nonparametric tests (e.g. Wilcoxon rank sums test) were used to compare treatment arms - Percent change of polyp counts from baseline to 6 months, ie [(6 months - baseline) x 100]/baseline (%). For each participant, first were matched polyps between baseline & 6 months by region and landmark and summed over all matched regions on number of polyps >2 mm to calculate total number of polyps >2 mm at baseline & 6 months, respectively. For participants refusing exit colonoscopy, 0% change entered as primary endpoint. Defined ITT All: All patients; if 6-month polyp counts missing = 0% change; ITT Measurable: All participants with baseline & 6 month polyp counts; ITT Evaluable: ITT Measurable participants who also took 80% of treatment, both overall as well as during final 60 days.
Time Frame: Baseline up to 6 months
Population: 112 patients were randomized to the study. Analysis was by intent to treat (ITT) with a total of 89 ITT participants measurable by having complete polyp information.
Measure: Mean (Standard Error); unit: percentage change in polyp count
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Number analyzed (Participants) | 55 | 57
percentage change in polyp count
  ITT All | -1 (0.11) | -11 (0.08)
  ITT Measurable | -1 (0.14) | -13 (0.10)
  ITT Evaluable | 10 (0.18) | -8 (0.12)

2. Primary Outcome: Number of Participants With Adverse Events Occurring at a Frequency of 5% or Grade 3 and Higher
Description: To determine the relative tolerability and safety of celecoxib + DFMO in FAP study participants. Includes only adverse events that occurred in at least 5% of the patients or a patient exhibited at least 1 grade 3 toxicity.
Time Frame: 6 months
Population: Total of 57 participants in Arm II, 1 participant is missing AE data
Measure: Count of Participants; unit: Participants
Groups:
- Arm I:Celecoxib, 400 mg p.o. BID Plus DFMO Placebo ( 60 Partic: Celecoxib, 400 mg p.o. BID plus DFMO placebo ( 60 participants with evaluable colon or rectum)
- Arm II: Celecoxib, 400 mg p.o. BID Plus DFMO 0.5 gm/m2/Day Rou: Celecoxib, 400 mg p.o. BID plus DFMO 0.5 gm/m2/day rounded down to the nearest 250mg dose ( 60 participants with evaluable colon or rectum). "
Arm/Group | Arm I:Celecoxib, 400 mg p.o. BID Plus DFMO Placebo ( 60 Partic | Arm II: Celecoxib, 400 mg p.o. BID Plus DFMO 0.5 gm/m2/Day Rou
Number analyzed (Participants) | 55 | 56
Participants
  High-frequency hearing loss | 4 | 7
  Fatigue | 11 | 3
  Diarrhoea | 6 | 4
  Heartburn/dyspepsia | 4 | 2
  Mucositis/stomatitis | 11 | 15
  Nausea/vomiting | 6 | 7
  Gout | 0 | 1
  Headache | 5 | 1

3. Secondary Outcome: Percentage Change in Global Colorectal Polyps Burden
Description: Percentage Change in Global Colorectal Polyps burden
Time Frame: 6 months
Population: A total of 89 participants had complete polyp information at baseline and 6 months.
Measure: Mean (Standard Error); unit: percentage change of total Polyps burden
Groups:
- Arm I: Celecoxib and Placebo: Celecoxib, 400 mg p.o. BID plus DFMO placebo ( 60 participants with evaluable colon or rectum)
- Arm II: Celecoxib and Eflornithine: Celecoxib, 400 mg p.o. BID plus DFMO 0.5 gm/m2/day rounded down to the nearest 250mg dose ( 60 participants with evaluable colon or rectum).
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Number analyzed (Participants) | 44 | 45
percentage change of total Polyps burden | -27 (6) | -40 (6)

4. Secondary Outcome: Percent Change in the Area of Plaque-like Duodenal Polyps
Time Frame: 6 months
Population: The data was inevaluable to determine the percent change in the area of plaque-like duodenal polyps
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Global Duodenal Polyp Burden
Time Frame: 6 months
Population: The data was inevaluable to determine the global duodenal polyp burden
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Percent Change in Polyp Size in Focal Area(s) of the Colorectum
Time Frame: Baseline up to 2 months after completion of study treatment
Population: No data collected to determine the percentage change in polyp size in focal area(s) of the colorectum.
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) collection was done monthly up to month 6 or early termination with all collected adverse events for randomized participants reported.
Description: Each adverse event (toxicity) reported counts once per participant. For example, if a participant had Grade 2 vomiting that increased to Grade 3 and then reduced to Grade 1 before going away, it counts as one event of Grade 3 vomiting.
Arm/Group | Arm I: Celecoxib and Placebo | Arm II: Celecoxib and Eflornithine
Serious Adverse Events (participants affected / at risk) | 0/55 | 3/57
Other Adverse Events (participants affected / at risk) | 53/55 | 48/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Celecoxib and Placebo (N=55) | Arm II: Celecoxib and Eflornithine (N=57)
Obstruction: Small Bowel NOS (Gastrointestinal disorders) | 0 | 1
Perforation GI - Colon (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Celecoxib and Placebo (N=55) | Arm II: Celecoxib and Eflornithine (N=57)
Allergies, seasonal (Immune system disorders) | 0 | 2
Allergic rhinitis (Immune system disorders) | 3 | 0
Allergic reaction (food) (Immune system disorders) | 0 | 1
High Frequency Hearing loss (Ear and labyrinth disorders) | 5 | 7
Otitis (Ear and labyrinth disorders) | 8 | 3
Tinnitus (Ear and labyrinth disorders) | 5 | 3
Hearing Impairment/Loss (Ear and labyrinth disorders) | 7 | 4
Hemoglobin Change (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Low Platelet (Blood and lymphatic system disorders) | 0 | 2
Cardiac ischemia (unstable angina) (Cardiac disorders) | 1 | 0
Chest tightness (Cardiac disorders) | 1 | 1
Hypertension (Cardiac disorders) | 3 | 1
Orthostatic Hypotension (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 2
Fatigue (General disorders) | 16 | 12
Fever (General disorders) | 1 | 2
Insomnia (General disorders) | 7 | 4
Night sweats (General disorders) | 0 | 1
Weight gain (General disorders) | 8 | 6
Weight loss (General disorders) | 1 | 2
Bruising (Skin and subcutaneous tissue disorders) | 3 | 3
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 2
Nodules (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 5 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash & Itching (Skin and subcutaneous tissue disorders) | 6 | 6
Other skin issues (Skin and subcutaneous tissue disorders) | 0 | 3
Hot flashes (Endocrine disorders) | 2 | 2
Anorexia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 4 | 3 — Burp, Distension/Bloating, Gas
Constipation (Gastrointestinal disorders) | 1 | 2
Dehydration (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 17 | 15
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1
Heartburn/Dyspepsia (Gastrointestinal disorders) | 14 | 11
Mucositis/Stomatitis (Gastrointestinal disorders) | 15 | 23
Nausea/Vomiting (Gastrointestinal disorders) | 12 | 16
Stricture: Rectum (Gastrointestinal disorders) | 0 | 1
Taste alteration (Gastrointestinal disorders) | 0 | 1
Ulcers (Gastrointestinal disorders) | 1 | 1 — Ileorectal Anastomosis, Rectum
Bloody stools (Blood and lymphatic system disorders) | 0 | 1
Hand & Wrist, Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 | 1
Hematuria (Blood and lymphatic system disorders) | 1 | 0
Nose Bleed (Blood and lymphatic system disorders) | 2 | 1
Rectum, Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 4 | 5
Vagina, Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 | 1
Cold Sore (mouth) (Infections and infestations) | 1 | 0
Conjunctiva (Infections and infestations) | 0 | 1
Ear Infection (Infections and infestations) | 0 | 1
Head & Nasal Infection (Infections and infestations) | 1 | 0
Head (fungus) Infection (Infections and infestations) | 1 | 0
Lung Infection (pneumonia) (Infections and infestations) | 1 | 0
Infection, Nose (yellow nasal drainage) (Infections and infestations) | 1 | 0
Infection, Right leg (spider bite) (Infections and infestations) | 0 | 1
Sinus Infection (Infections and infestations) | 1 | 0
Infection, Stomach (Infections and infestations) | 2 | 3
Infection, Ungual (Infections and infestations) | 0 | 2
Infection, Upper airway NOS (Infections and infestations) | 3 | 3
Edema (Blood and lymphatic system disorders) | 4 | 6
ALT, SGPT Changes (Metabolism and nutrition disorders) | 1 | 1
AST, SGOT Changes (Metabolism and nutrition disorders) | 0 | 1
Alkaline phosphatase Changes (Metabolism and nutrition disorders) | 1 | 0
Creatinine Changes (Metabolism and nutrition disorders) | 0 | 1
Elevated LDL (Metabolism and nutrition disorders) | 0 | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 | 0
Hypercholestremia & Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Proteinuria (Metabolism and nutrition disorders) | 1 | 1
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 | 2 — Gait and standing
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle/bone soreness from fall (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw tightness (left side) (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower jaw tear (Musculoskeletal and connective tissue disorders) | 0 | 1
Puncture wound (Musculoskeletal and connective tissue disorders) | 0 | 1
Sutures in shoulder (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive Disturbance (ADD) (Nervous system disorders) | 1 | 0 — Neurology
Dizziness (Nervous system disorders) | 7 | 6
Memory Impairment (Nervous system disorders) | 1 | 1
Mood Alteration : Anxiety (Nervous system disorders) | 2 | 0
Mood alteration : Depression (Nervous system disorders) | 1 | 1
Numbness (Nervous system disorders) | 3 | 2
Numbness & Tingling (Nervous system disorders) | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Tingling (Nervous system disorders) | 0 | 1
Blurred Vision (Eye disorders) | 3 | 1 — Ocular/Visual
Bright lights (Eye disorders) | 1 | 0
Decreased vision (left eye) (Eye disorders) | 1 | 0
Decreased visual acuity (Eye disorders) | 1 | 0
Dry eye syndrome (Eye disorders) | 0 | 1
Eyelid scratch (Eye disorders) | 1 | 0
Near sighted (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Tired eyes (Eye disorders) | 1 | 0
Unequal pupils (Eye disorders) | 1 | 0
Vision-floaters (Eye disorders) | 0 | 1
Watery eye (Eye disorders) | 0 | 1
Yellow discoloration (right ey (Eye disorders) | 0 | 1
Pain, Abdomen (General disorders) | 14 | 9 — Pain
Pain, Wrist, Arm & Shoulder (General disorders) | 2 | 2
Pain, Back (General disorders) | 5 | 4 — Flank and sides
Pain, Breast (tenderness) (General disorders) | 0 | 1
Pain, Breast bone (General disorders) | 0 | 1
Pain, Cardiac/Heart (General disorders) | 1 | 1
Pain, Chest/thorax NOS (General disorders) | 1 | 1
Pain, Ear (General disorders) | 2 | 3
Pain, Extremity-limb (General disorders) | 2 | 0
Pain, Groin/Loin/Thigh (General disorders) | 1 | 2
Headache (General disorders) | 16 | 14
Pain, Joint/Musculoskeletal (General disorders) | 6 | 2
Pain, Muscle (General disorders) | 4 | 2
Pain, Neck (General disorders) | 1 | 0
Pain, Oral-gums (General disorders) | 1 | 0
Pain, Rectum (General disorders) | 2 | 1
Pain, Throat/Pharynx (General disorders) | 1 | 6
Pain, Vagina (cramping) (General disorders) | 0 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 0 — Pulmonary/Upper Respiratory
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Burning with urination (Renal and urinary disorders) | 0 | 1
Crystals in urine (Renal and urinary disorders) | 1 | 0
Kidney stone (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 1 | 0
Irritation around genitals (Reproductive system and breast disorders) | 1 | 0
Intra-Operative Injury Extremity-Upper (Injury, poisoning and procedural complications) | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Following reports of COX-2 inhibitor-associated cardiovascular toxicities, trial suspended from December 17, 2004 to March 18, 2005 pending reevaluation of cardiovascular risks, only two sites resumed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less